CLINICAL TRIAL: NCT04354571
Title: Evaluation of Post Operative Analgesia of the Erector Spinae Plane Block in Pediatric Patients Undergoing Hip Surgery: a Randomized Control Trial
Brief Title: Erector Spinae Plane Block in Pediatric Hip Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Yasser Mohamed Mohamed Osman, assistant professor of anesthesia Alexandria university, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1234
Record Dates: First submitted 2020-04-12; First posted 2020-04-21 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: closed envelope technique
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP (Erector spinae block): (Experimental): were given general anesthesia plus Erector spinae plane block
  Interventions: Procedure: Erector spinae plane block
- GROUP (caudal block): (Active Comparator): were given general anesthesia plus caudal block
  Interventions: Procedure: caudal block

INTERVENTIONS:
Procedure: Erector spinae plane block — An ultrasound-guided Erector spinae plane block was performed with the patient lying on the his side and the surgical side on the top. After skin disinfection, sterile draping was be placed and the ultrasound probe was sheathed. The level of the block was the transverse process of L2. The block was performed using a 9-12 MHz linear probe (LOGIQe, GE Healthcare, USA), which was placed in a parasagittal plane 1 cm from the posterior midline. The deep plane to the erector spinae muscle (ESM) was identified, and a 22 G, 50 mm insulated needle (Sonoplex Stim, Pajunk, Germany) was inserted cranio-caudally in plane between the transverse process and the fascia of the ESM. After negative aspiration, 0.3 ml/kg of 0.25% bupivacaine was injected to confirm the correct position by visualizing the solution lifting the ESM off the transverse process.
  Arms: GROUP (Erector spinae block):
Procedure: caudal block — caudal block was performed using anatomical landmarks and ultrasound guided and confirmed with a concentration of bupivacaine of 0.25%.
  Arms: GROUP (caudal block):

SUMMARY:
Hip Surgery in pediatric patients is considered an extremely painful procedure. Managing pain in this surgery is challenging even with several available options, each with limitations. Erector spinae plane (ESP) block is a novel technique that has been used in different types of surgery, with promising results. Many case reports for use of ESPB are available in the literature but to our knowledge, no cohort studies or randomized controlled trials have been performed on ESPB for hip surgery in pediatrics age group against a traditional method as caudal block.1,2 AIM OF WORK

. The Primary outcome of this study is to compare the efficacy of analgesia resulting from the Erector spinae plane block versus the caudal block in pediatric patients undergoing hip surgery using the FLACC score and the duration of the analgesia of both methods till the first rescue analgesic.

The Secondary outcome is to compare the analgesic rescue frequency and total dose given in both groups as well as comparing the complications that might occur from each analgesic technique.

ELIGIBILITY:
Inclusion Criteria:

* ASA I II scheduled for hip surgery.

Exclusion Criteria:

* • Parent refusal

  * Coagulopathy
  * Patient with congenital heart disease
  * Infection at the site of puncture
  * Significant spinal anatomical anomaly
  * Patient with neuromuscular disorder
  * Any known allergy to the drug used

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2019-08-11 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | 1 day .
  Pain was assessed using face, legs, activity, and cry consolability scale [FLACC] 1-10 1 is no pain and 10 is the worst pain.

SECONDARY OUTCOMES:
complications | through study completion, an average of 1 day
  not any complication related to the block

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No